CLINICAL TRIAL: NCT06206447
Title: Comparison of Short-term Application of Dialysis Catheter With Tunnel-cuffed Catheter Versus Non-ccuffed Catheter: a Multicenter Prospective Cohort Study
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Beijing Friendship Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: BFHHZML20230013
Record Dates: First submitted 2024-01-04; First posted 2024-01-16 (Actual); Last update posted 2024-01-16 (Actual); Status verified 2023-10

CONDITIONS: Clarify the Difference of Short-term Infection Rate Between Diffrent Catheter

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Tunnel-cuffed Catheter Group: Hemodialysis patient with Tunnel-cuffed Catheter in right internal jugular vein
  Interventions: Procedure: Tunnel-cuffed Catheter
- Non-ccuffed Catheter Group: Hemodialysis patient with Non-cuffed Catheter in right internal jugular vein
  Interventions: Procedure: Non-ccuffed Catheter

INTERVENTIONS:
Procedure: Tunnel-cuffed Catheter — Tunnel-cuffed Catheter in right internal jugular vein
  Groups: Tunnel-cuffed Catheter Group
Procedure: Non-ccuffed Catheter — Non-ccuffed Catheter in right internal jugular vein
  Groups: Non-ccuffed Catheter Group

SUMMARY:
Through a multi-center, prospective cohort study, hemodialysis patients with right internal jugular vein catheterization were collected and divided into tunnel-cuffed catheter group and non-cuffed catheter group according to the types of catheterization. The incidence of catheter infection, thrombosis and other complications between the two groups were compared.To clarify the difference of short-term infection rate between tunnel-cuffed catheter and non-cuffed catheter.

ELIGIBILITY:
Inclusion Criteria:

* ① Age ≥18 years; ② Uremia, clinical evaluation needs to start hemodialysis immediately, and the right internal jugular vein catheterization is the vascular access for the subjects. ③ Subjects who underwent right internal jugular vein catheterization on regular hemodialysis due to poor internal fistula function and the recovery time of internal fistula was ≥4 weeks; ④ Patients with AKI who need renal replacement therapy and underwent catheterization in the right internal jugular vein, and the renal replacement time is ≥4 weeks.

Exclusion Criteria:

* ① Subjects with previous history of central venous thrombosis, stenosis, infection, etc. ② The subjects were not dialyzed three times a week; ③ Other subjects with central venous catheterization, including left internal jugular vein, femoral vein and subclavian vein; ④ Those who take immunosuppression for a long time.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patient who needs hemodialysis with catheter in right internal jugular vein
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2023-11-01 (Actual); Primary Completion 2025-10-31 (Estimated); Study Completion 2025-10-31 (Estimated)

PRIMARY OUTCOMES:
Cumulative incidence of catheter infection within 3 months after catheterization | within 3 months after catheterization
  Cumulative incidence of catheter infection within 3 months after catheterization

SECONDARY OUTCOMES:
Cumulative incidence of catheter infection within 2 months after catheterization | within 2 months after catheterization
  Cumulative incidence of catheter infection within 2 months after catheterization
Cumulative incidence of catheter infection within 1 months after catheterization | within 1 months after catheterization
  Cumulative incidence of catheter infection within 1 months after catheterization

OTHER OUTCOMES:
The incidence of catheter dysfunction | within 3 months after catheterization
  The incidence of catheter dysfunction

CONTACTS AND LOCATIONS:
Locations (1):
- Beijing Friedship Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided